CLINICAL TRIAL: NCT02972905
Title: A Single Center, Double-blind, Randomized, Placebo-controlled, Parallel, Single and Repeat, Dose-ascending Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GSK2269557 Administered Via the ELLIPTA™ Dry Powder Inhaler to Healthy Japanese Subjects
Brief Title: Study to Evaluate Safety, Tolerability and Pharmacokinetics of GSK2269557 to Japanese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205759
Record Dates: First submitted 2016-10-14; First posted 2016-11-25 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: pharmacokinetics; GSK2269557; Dry powder Inhaler (DPI); tolerability; safety; ELLIPTA
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Session 1: Placebo (Placebo Comparator): Subjects will receive a single dose inhalation of GSK2269557 matching placebo via the ELLIPTA DPI. The washout period between the two dosing sessions will be at least 10 days.
  Interventions: Drug: Placebo ELLIPTA DPI
- Session 1: GSK2269557 200 mcg (Experimental): Subjects will receive a single dose inhalation of GSK2269557 200 mcg via the ELLIPTA DPI. The washout period between the two dosing sessions will be at least 10 days.
  Interventions: Drug: GSK2269557 ELLIPTA DPI
- Session 1: GSK2269557 500 mcg (Experimental): Subjects will receive a single dose inhalation of GSK2269557 500 mcg via the ELLIPTA DPI. The washout period between the two dosing sessions will be at least 10 days.
  Interventions: Drug: GSK2269557 ELLIPTA DPI
- Session 1: GSK2269557 700 mcg (Experimental): Subjects will receive a single dose inhalation of GSK2269557 700 mcg via the ELLIPTA DPI. The washout period between the two dosing sessions will be at least 10 days.
  Interventions: Drug: GSK2269557 ELLIPTA DPI
- Session 2: Placebo (Placebo Comparator): Subjects will receive repeated doses of GSK2269557 matching Placebo once daily via the ELLIPTA DPI for 10 days. The washout period between the two dosing sessions will be at least 10 days.
  Interventions: Drug: Placebo ELLIPTA DPI
- Session 2: GSK2269557 200 mcg (Experimental): Subjects will receive repeated doses of GSK2269577 200mcg once daily via the ELLIPTA DPI for 10 days. The washout period between the two dosing sessions will be at least 10 days.
  Interventions: Drug: GSK2269557 ELLIPTA DPI
- Session 2: GSK2269557 500 mcg (Experimental): Subjects will receive repeated doses of GSK2269577 500mcg once daily via the ELLIPTA DPI for 10 days. The washout period between the two dosing sessions will be at least 10 days.
  Interventions: Drug: GSK2269557 ELLIPTA DPI
- Session 2: GSK2269557 700 mcg (Experimental): Subjects will receive repeated doses of GSK2269577 700mcg once daily via the ELLIPTA DPI for 10 days. The washout period between the two dosing sessions will be at least 10 days.
  Interventions: Drug: GSK2269557 ELLIPTA DPI

INTERVENTIONS:
Drug: GSK2269557 ELLIPTA DPI — GSK2269557 ELLIPTA DPI contains GSK2269557 blended with lactose and magnesium stearate. This will be supplied in two strength of 100 mcg per blister and 500 mcg per blister.
  Arms: Session 1: GSK2269557 200 mcg; Session 1: GSK2269557 500 mcg; Session 1: GSK2269557 700 mcg; Session 2: GSK2269557 200 mcg; Session 2: GSK2269557 500 mcg; Session 2: GSK2269557 700 mcg
Drug: Placebo ELLIPTA DPI — Placebo ELLIPTA DPI contains lactose
  Arms: Session 1: Placebo; Session 2: Placebo

SUMMARY:
GSK2269557 is a potent and highly selective inhaled Phosphoinositide 3-Kinase (PI3K) delta inhibitor being developed as an anti-inflammatory and anti-infective agent for the treatment of inflammatory airway diseases, such as chronic obstructive pulmonary disease (COPD). The purpose of the study is to assess the safety, tolerability and pharmacokinetics (PK) of single and repeat doses of GSK2269557 administered via the ELLIPTA dry powder inhaler (DPI) to healthy Japanese subjects. This is the first time for Japanese subjects that GSK2269557 will be administered via the ELLIPTA DPI with the addition of magnesium stearate.

In each group of this study, subjects will receive a single dose of either GSK2269557 or placebo in Session 1 and receive daily dose of GSK2269557 or placebo for 10 days in Session 2. Session 1 of the next dose strength may be run in parallel with the Session 2 of the previous dose. The doses planned for the study are 200 micrograms (mcg), 500 mcg and 700 mcg. There will be at least 10 days washout between the two dosing sessions. Follow up period will start 10 days (+-1 day) after the last dose of Session 2. A total number of 36 subjects will be enrolled for the study with 27 subjects receiving a dose strength of GSK2269557 and 9 subjects will receive each dose strength of GSK2269557. ELLIPTA is a trademark of the GSK group of companies.

ELIGIBILITY:
Inclusion Criteria

* Participant must be 20 to 64 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and ECG. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Normal spirometry (forced expiratory volume in 1 second >=80% of predicted) at Screening.
* Body weight >=50 kilograms (kg) and body mass index (BMI) within the range 18.5 to 24.9 kg/square meter (m^2) (inclusive).
* Japanese Male: A male participant must agree to use contraception of this protocol during the treatment period and until follow up visit.
* Capable of giving signed informed consent as described in restrictions listed in the informed consent form (ICF).

Exclusion Criteria

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data
* Abnormal blood pressure as determined by the investigator
* ALT >1.5x upper limit of normal (ULN)
* Bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* QTcF >450 milliseconds (msec).
* Past or intended use of over-the-counter or prescription medication including herbal medications within 14 days prior to dosing.
* History of donation of blood or blood products >=400 milliliters (mL) within 3 months or >=200 mL within 1 month prior to screening
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day
* Current enrollment or past participation within the last 30 days before signing of consent in this clinical study involving an investigational study treatment or any other type of medical research
* The subject is positive Serological test for syphilis (rapid plasma reagin and Treponema pallidum), Human immunodeficiency virus (HIV) Antigen/Antibody, Hepatitis B surface antigen (HbsAg), Hepatitis C virus (HCV) antibody, or Human T-cell lymphotropic virus type 1 (HTLV-1) antibody at screening.
* Positive pre-study drug screen
* Regular use of known drugs of abuse
* Regular alcohol consumption within 6 months prior to the study defined as: for an average weekly intake of >14 units for males. One unit is equivalent to 350 ml of beer, 150 ml of wine or 45 ml of 80 proof distilled spirits
* Smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening
* Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with any adverse event(s) (AE) and serious adverse event(s) (SAE) | Approximately up to 37 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in persisting disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment will be categorized as SAE.
Session 1: Number of subjects having abnormal clinical laboratory parameters as a measure of safety | Approximately up to 4 days
  Blood samples will be collected to analyse blood urea nitrogen, creatinine, glucose (fasting), uric acid, high density lipoprotein-cholesterol, amylase, potassium, sodium, calcium, triglycerides, lactate dehydrogenase (LDH), chloride, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), total cholesterol, gamma-glutamyl transpeptidase (GGT), phosphorus, total bilirubin, direct bilirubin, total protein, albumin, low density lipoprotein-cholesterol, creatine phosphokinase (CPK)
Session 2: Number of subjects having abnormal clinical laboratory parameters as a measure of safety | Approximately up to 22 days
  Blood samples will be collected to analyse blood urea nitrogen, creatinine, glucose (fasting), uric acid, high density lipoprotein-cholesterol, amylase, potassium, sodium, calcium, triglycerides, LDH, chloride, AST, ALT, ALP, total cholesterol, GGT, phosphorus, total bilirubin, direct bilirubin, total protein, albumin, low density lipoprotein-cholesterol, CPK
Session 1:Number of subjects having abnormal hematology laboratory parameters as a measure of safety | Approximately up to 4 days
  Blood samples will be collected to analyse platelet count, Red Blood Cells (RBC) count, hemoglobin, hematocrit, RBC Indices, mean corpuscular volume ( MCV), mean corpuscular hemoglobin (MCH), percent reticulocytes, White Blood Cells (WBC), neutrophils, lymphocytes, monocytes, eosionophils, and basophils
Session 2: Number of subjects having abnormal hematology laboratory parameters as a measure of safety | Approximately up to 22 days
  Blood samples will be collected to analyse platelet count, RBC count, hemoglobin, hematocrit, RBC Indices, MCV, MCH, percent reticulocytes, WBC, neutrophils, lymphocytes, monocytes, eosionophils, and basophils
Session 1: Number of subjects having abnormal urinalysis as a measure of safety | Approximately up to 4 days
  Urine samples will be collected to analyse specific gravity, pH, glucose, protein, blood, ketones, bilirubin, and urobilinogen for dipstick, and microscopic examination
Session 2: Number of subjects having abnormal urinalysis as a measure of safety | Approximately up to 22 days
  Urine samples will be collected to analyse specific gravity, pH, glucose, protein, blood, ketones, bilirubin, and urobilinogen for dipstick, and microscopic examination
Session 1: Body temperature assessment as a safety measure | Approximately up to 4 days
  Temperature will be recorded in a supine position after 5 minutes rest
Session 2: Body temperature assessment as a safety measure | Approximately up to 22 days
  Temperature will be recorded in a supine position after 5 minutes rest
Session 1: Blood pressure assessment as a safety measure | Approximately up to 4 days
  Systolic and diastolic blood pressure will be measured in a supine positon after 5 minutes rest
Session 2: Blood pressure assessment as a safety measure | Approximately up to 22 days
  Systolic and diastolic blood pressure will be measured in a supine position after 5 minutes rest
Session 1: Measurement of pulse rate as a safety measure | Approximately up to 4 days
  Pulse rate will be measured in a supine position after 5 minutes rest
Session 2: Measurement of pulse rate as a safety measure | Approximately up to 22 days
  Pulse rate will be measured in a supine position after 5 minutes rest
Session 1: Electrocardiogram (ECG) assessment as a measure of safety. | Approximately up to 4 days
  Single 12-lead ECG will be obtained in a supine position after 5 minutes rest using an ECG machine that measures PR, QRS, QT, and Corrected QT interval by Fridericia's formula (QTcF) intervals. Single ECGs will be obtained at each time point.
Session 2: ECG assessment as a measure of safety. | Approximately up to 22 days
  Single 12-lead ECG will be obtained in a supine position after 5 minutes rest using an ECG machine that measures PR, QRS, QT, and QTcF intervals. Single ECGs will be obtained at each time point.
Session 1: Spirometry assessment as a safety measure | Approximately up to 4 days
  Spirometry assessments will be performed whilst the subject is in a standing position. Assessments will be repeated until 3 technically acceptable measurements have been made.
Session 2: Spirometry assessment as a safety measure | Approximately up to 22 days
  Spirometry assessments will be performed whilst the subject is in a standing position. Assessments will be repeated until 3 technically acceptable measurements have been made.
Session 1: Area under the plasma concentration curve (AUC) from time zero to the time of last quantifiable concentration [AUC(0-t)] | Pre-dose, 5, 15, 30 minutes (min), 1, 2 , 4 , 6, 12, 24, 36, 48, and 72hours (h) post-dose
  Blood samples will be collected at pre-dose and at specific post dose time points for calculating AUC [0-t]
Session 1: AUC from time zero to 24 hours post dose [AUC(0-24)] of GSK2269557 following a single dose administration | Pre-dose, 5, 15, 30 min, 1, 2 , 4 , 6, 12, 24, 36, 48, and 72h post-dose
  Blood samples will be collected at pre-dose and at specific post dose time points for calculating AUC[0-24]
Session 1: AUC from time zero to infinity [AUC(0-infinity)] of GSK2269557 following a single dose administration | Pre-dose, 5, 15, 30 min, 1, 2 , 4 , 6, 12, 24, 36, 48, and 72h post-dose
  Blood samples will be collected at pre-dose and at specific post dose time points for calculating AUC (0-infinity).
Session 2: AUC from time zero to the time of last quantifiable concentration [AUC(0-t)] of GSK2269557 following repeat dose administration | Day 1: pre-dose, 5 min and 24 h post-dose; Day 2: 5 min post-dose; Days 3, 4, 5, 6, 7, 8, and 9: pre-dose and 5 min post-dose; Day 10: pre-dose, and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h post-dose; 24 h, 48 h, 72 h, 96 h and 120 h post-Day 10 dose
  Blood samples will be collected at pre-dose and at specific post dose time points for calculating AUC [0-t]
Session 2: AUC from time zero to 24 hours post dose [AUC(0-24)] of GSK2269557 following repeat dose administration | Day 1: pre-dose, 5 min and 24 h post-dose; Day 2: 5 min post-dose; Days 3, 4, 5, 6, 7, 8, and 9: pre-dose and 5 min post-dose; Day 10: pre-dose, and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h post-dose; 24 h, 48 h, 72 h, 96 h and 120 h post-Day 10 dose
  Blood samples will be collected at pre-dose and at specific post dose time points for calculating AUC[0-24]
Session 2: AUC from time zero to infinity [AUC(0-infinity)] of GSK2269557 following repeat dose administration | Day 1: pre-dose, 5 min and 24 h post-dose; Day 2: 5 min post-dose; Days 3, 4, 5, 6, 7, 8, and 9: pre-dose and 5 min post-dose; Day 10: pre-dose, and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h post-dose; 24 h, 48 h, 72 h, 96 h and 120 h post-Day 10 dose
  Blood samples will be collected at pre-dose and at specific post dose time points for calculating AUC (0-infinity)
Session 1: Trough observed plasma drug concentration (Ctrough) of GSK2269557 following a single dose administration | Pre-dose, 5, 15, 30 minutes (min), 1, 2 , 4 , 6, 12, 24, 36, 48, and 72h post-dose
  Blood samples will be collected at pre-dose and at specific post dose time points for calculating Ctrough
Session 1: Maximum observed plasma concentration (Cmax) of GSK2269557 following a single dose administration | Pre-dose, 5, 15, 30 minutes (min), 1, 2 , 4 , 6, 12, 24, 36, 48, and 72h post-dose
  Blood samples will be collected at pre-dose and at specific post dose time points for calculating Cmax
Session 1: Maximum/trough observed plasma drug concentration (Cmax/Ctrough) of GSK2269557 following a single dose administration | Pre-dose, 5, 15, 30 minutes (min), 1, 2 , 4 , 6, 12, 24, 36, 48, and 72h post-dose
  Blood samples will be collected at pre-dose and at specific post dose time points for calculating Cmax/Ctrough
Session 2: Trough observed plasma drug concentration (Ctrough) of GSK2269557 following repeat dose administration | Day 1: pre-dose, 5 min and 24 h post-dose; Day 2: 5 min post-dose; Days 3, 4, 5, 6, 7, 8, and 9: pre-dose and 5 min post-dose; Day 10: pre-dose, and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h post-dose; 24 h, 48 h, 72 h, 96 h and 120 h post-Day 10 dose
  Blood samples will be collected at pre-dose and at specific post dose time points for calculating Ctrough
Session 2: Maximum observed plasma concentration (Cmax) of GSK2269557 following repeat dose administration | Day 1: pre-dose, 5 min and 24 h post-dose; Day 2: 5 min post-dose; Days 3, 4, 5, 6, 7, 8, and 9: pre-dose and 5 min post-dose; Day 10: pre-dose, and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h post-dose; 24 h, 48 h, 72 h, 96 h and 120 h post-Day 10 dose
  Blood samples will be collected at pre-dose and at specific post dose time points for calculating Cmax
Session 2: Maximum/trough observed plasma drug concentration (Cmax/Ctrough) of GSK2269557 following repeat dose administration | Day 1: pre-dose, 5 min and 24 h post-dose; Day 2: 5 min post-dose; Days 3, 4, 5, 6, 7, 8, and 9: pre-dose and 5 min post-dose; Day 10: pre-dose, and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h post-dose; 24 h, 48 h, 72 h, 96 h and 120 h post-Day 10 dose
  Blood samples will be collected at pre-dose and at specific post dose time points for calculating Cmax/Ctrough
Session 1: Time to maximum observed plasma drug concentration (Tmax) of GSK2269557 following a single dose administration | Pre-dose, 5, 15, 30 min, 1, 2 , 4 , 6, 12, 24, 36, 48, and 72h post-dose
  Blood samples will be collected at pre-dose and at specific post dose time points for calculating tmax
Session 1: Terminal half-life (t1/2) of GSK2269557 following a single dose administration | Pre-dose, 5, 15, 30 min, 1, 2 , 4 , 6, 12, 24, 36, 48, and 72h post-dose
  Blood samples will be collected at pre-dose and at specific post dose time points for calculating t1/2
Session 2: Time to maximum observed plasma drug concentration (Tmax) of GSK2269557 following repeat dose administration | Day 1: pre-dose, 5 min and 24 h post-dose; Day 2: 5 min post-dose; Days 3, 4, 5, 6, 7, 8, and 9: pre-dose and 5 min post-dose; Day 10: pre-dose, and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h post-dose; 24 h, 48 h, 72 h, 96 h and 120 h post-Day 10 dose
  Blood samples will be collected at pre-dose and at specific post dose time points for calculating tmax
Session 2: Terminal half-life (t1/2) of GSK2269557 following repeat dose administration | Day 1: pre-dose, 5 min and 24 h post-dose; Day 2: 5 min post-dose; Days 3, 4, 5, 6, 7, 8, and 9: pre-dose and 5 min post-dose; Day 10: pre-dose, and 5 min, 30 min, 1 h, 2 h, 4 h, 6 h post-dose; 24 h, 48 h, 72 h, 96 h and 120 h post-Day 10 dose
  Blood samples will be collected at pre-dose and at specific post dose time points for calculating tmax and t1/2
Ratio of accumulation factor (Ro) of GSK2269557 following single and repeat inhalations | Day 1 of session 2 and day 10 of session 2
  Ro is defined as AUC(0-24) of Session 2 at day10 divided by AUC(0-24) of Session1
Ratio of accumulation factor (Rs) of GSK2269557 following single and repeat inhalations | Day 1 of session 2 and day 10 of session 2
  Rs is defined as AUC(0-24) of Session 2 at day10 divided by AUC(0-infinity) of Session 1
Ratio of accumulation factor (R[Cmax]) of GSK2269557 following single and repeat inhalations | Day 1 of session 2 and day 10 of session 2
  R[Cmax] is defined as Cmax of Session 2 at day10 divided by Cmax of Session 1
Ratio of accumulation factor (R[Ctrough]) of GSK2269557 following single and repeat inhalations | Day 1 of session 2 and day 10 of session 2
  R[Ctrough] is defined as Ctrough of Session 2 at day10 divided by C24 of Session 1

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fukuoka, Japan